CLINICAL TRIAL: NCT03363997
Title: A Randomized, Open-label Trial to Evaluate the Pharmacokinetics and Pharmacodynamics of 3 Dosages of Estriol After Continuous Vaginal Administration for 21 Days in Healthy, Post-menopausal Women
Brief Title: Pharmacokinetics and Pharmacodynamics of 3 Dosages of Estriol After Continuous Vaginal Administration for 21 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: SocraTec R&D GmbH (Other)
Responsible Party: Principal Investigator, Gilberto De Nucci, Doctor, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDN 005/16
Record Dates: First submitted 2017-11-27; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Menopause
Keywords: estriol; pharmacokinetic; pharmacodynamic; hormone replacement therapy; vaginal ring administration
MeSH Terms: interventions — Estriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test 1 vaginal ring (Experimental): Single vaginal application of 1 vaginal ring containing 100 mg estriol, with delivery rate of 0.125 mg/day over 21 days
  Interventions: Drug: Estriol 0.125 mg/day
- Test 2 vaginal ring (Experimental): Single vaginal application of 1 vaginal ring containing 300 mg estriol, with delivery rate of 0.250 mg/day over 21 days
  Interventions: Drug: Estriol 0.250 mg/day
- Test 3 vaginal ring (Experimental): Single vaginal application of 1 vaginal ring containing 600 mg estriol, with delivery rate of 0.500 mg/day over 21 days
  Interventions: Drug: Estriol 0.500 mg/day

INTERVENTIONS:
Drug: Estriol 0.125 mg/day — Application of one vaginal ring
  Arms: Test 1 vaginal ring
Drug: Estriol 0.250 mg/day — Application of one vaginal ring
  Arms: Test 2 vaginal ring
Drug: Estriol 0.500 mg/day — Application of one vaginal ring
  Arms: Test 3 vaginal ring

SUMMARY:
This clinical trial evaluated the pharmacokinetics and pharmacodynamics of estriol in healthy post-menopausal women after the application of one vaginal ring containing one of three different dosages of estriol (100 mg (Test 1), 300 mg (Test 2) or 600 mg (Test 3)) with continuous delivery (0.125, 0.250 or 0.500 mg/day) for 21 days. And also, characterized its safety and tolerability.

DETAILED DESCRIPTION:
This phase I, single center, open-label, randomised (allocation to treatment), balanced, single dose trial was performed in a parallel-group design. The subjects were randomly assigned to one of the 3 possible treatments (single vaginal application of 1 vaginal ring containing 100, 300 or 600 mg estriol, with delivery rate of 0.125, 0.250 or 0.500 mg/day over 21 days.

Blood samples were collected at 0.5 h prior to drug application, 1, 2, 4, 6, 12, 24, 48, 96, 144, 216, 288, 360, 432 h after application; 5 min prior to removal, i.e., 21 d after application (study day 22), as well as 6, 12 and 24 h after removal to characterise pharmacokinetic parameters of estriol in plasma.

Serum concentrations of follicle stimulating hormone (FSH), luteinising hormone (LH) and sex hormone binding globulin (SHBG) and gynaecological parameters (cytology of vaginal smear, the maturation index and the vaginal pH) were evaluated as pharmacodynamic parameters.

The safety and tolerability was assessed by endometrial thickness and documentation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index (BMI) ≥18.5 kg/m² and ≤ 30.0 kg/m²
* Postmenopausal state: FSH (plasma) ≥ 40 IU/l, estradiol (serum) ≤ 20 pg/ml last spontaneous menstruation at least 12 months ago
* Normal transvaginal endometrial scan (endometrial thickness < 5 mm)
* Good state of health
* Non-smoker or ex-smoker for at least 6 month
* Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

* Existing cardiac, hepatic and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability and/or pharmacokinetics and/or pharmacodynamics of the active ingredient
* History of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
* Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
* Subjects with severe allergies or multiple drug allergies, unless it is judged as not relevant for the clinical trial by the investigator
* Positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test (if positive to be verified by test for HBc-IgM) or anti-HCV-test
* Presence or history of venous or arterial thrombosis (e.g. deep venous thrombosis, pulmonary embolism)
* Known, past or suspected breast cancer or increased familiar risk for development
* Known or suspected estrogen-dependent malignant tumours (e.g. endometrial or breast cancer)
* Undiagnosed genital bleeding
* Acute vaginal infection or other diseases prohibiting the placement of vaginal ring
* History of endometrial hyperplasia
* Migraine or frequent episodes of severe headache
* History of or current drug or alcohol dependence
* Subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
* Regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
* Blood donation or other blood loss of more than 400 ml within the last 3 months prior to individual enrolment of the subject
* Participation in a clinical trial during the last 6 months prior to individual enrolment of the subject
* Concomitant systemic therapy with antibiotics, which might interfere with enterohepatic recirculation (e.g. cephalosporines, neomycin, ampicillin or tetracyclines)
* Use of sex hormones within 6 months (oral, transdermal, vaginal) or 8 months (intramuscular administered depot preparations used once per month) or 12 months (intramuscular administered depot preparations used once per 3 months) before screening
* Use of systemic or topical medications or substances which oppose the study objectives or which might influence them within 8 weeks before screening examination
* Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Measurement of estriol plasma levels | 0-22 days
  Blood sampling for the determination of plasma levels of estriol in participants of each treatment group.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of estriol | 0-22 days
  Determination of Cmax for estriol based on plasma concentrations of samples obtained.
Area Under the Curve (AUC) for estriol | 0-22 days
  Calculation of the AUC for estriol based on plasma concentrations of samples obtained.
Characterisation of follicle stimulating hormone (FSH) | 0-22 days
  Determination of serum concentrations of FSH under the three treatments
Characterisation of luteinising hormone (LH) | 0-22 days
  Determination of serum concentrations of LH under the three treatments
Characterisation of sex hormone binding globulin (SHBG) | 0-22 days
  Determination of serum concentrations of SHBG under the three treatments
Characterisation of cytology of vaginal smear | 0-22 days
  Characterisation of cytology of vaginal smear (parabasal, intermediate and superficial cells) under the three treatments
Calculation of maturation index | 0-22 days
  Calculation of maturation index under the three treatments
Determination of vaginal pH | 0-22 days
  Determination of vaginal pH under the three treatments
Number of adverse events per participant | up to 22days after treatment
  Number of adverse events, in each treatment group, including clinically relevant alterations of vital signs and laboratory tests results.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, MD, Principal Investigator — Galeno Desenvolvimento de Pesquisas Clinicas Ltda
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252